CLINICAL TRIAL: NCT02128464
Title: Comparison of Customized Cutting Block (Visionaire™) and Conventional Total Knee Arthroplasty: A Prospective Randomized Control Trial
Brief Title: Outcome of TKA Using Customized Cutting Block Compared With Conventional Intramedullary Cutting Guide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Phonthakorn Panichkul, Phonthakorn Panichkul, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OrthoTu-02; OrthoTu-02 (Other: Thammasat University)
Record Dates: First submitted 2013-11-25; First posted 2014-05-01 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Total Knee Arthroplasty; Customized Cutting Block; Conventional Intramedullary Cutting Guide
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard knee cutting guides (Active Comparator): Standard cutting guides use traditional instrumentation to determine knee implant positions. During surgery, a rod is placed in the leg bone and the cutting guide is attached to that rod.
  Interventions: Procedure: Standard knee cutting guides
- Patient specific cutting guides (Active Comparator): Patient specific cutting guides are custom-made for each patient based on Magnetic Resonance Imaging (MRI). Before surgery, MRI of the knee is done and used to create a cutting guide that is formed to the exact shape of the knee. The patient specific cutting guides have platforms that can be attached to the bone, so the rod does not need to be placed in the leg bone.
  Interventions: Procedure: Patient specific cutting guides

INTERVENTIONS:
Procedure: Patient specific cutting guides — Patient specific cutting guides are custom-made for each patient based on Magnetic Resonance Imaging (MRI). Before surgery, MRI of the knee is done and used to create a cutting guide that is formed to the exact shape of the knee. The patient specific cutting guides have platforms that can be attached to the bone, so the rod does not need to be placed in the leg bone.
  Arms: Patient specific cutting guides
Procedure: Standard knee cutting guides — Standard cutting guides use traditional instrumentation to determine knee implant positions. During surgery, a rod is placed in the leg bone and the cutting guide is attached to that rod.
  Arms: Standard knee cutting guides

SUMMARY:
Customized cutting block and conventional cutting guide are both effective in improving accuracy and function of OA knee patients.

DETAILED DESCRIPTION:
Customized cutting block and conventional cutting guide are both effective in improving accuracy and function of osteoarthritic knee patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-90
* Diagnosis of osteoarthritis or rheumatoid arthritis of the knee and qualify for surgery, as indicated by one of the following:
* Painful and disabled knee joint resulting from osteoarthritis where one or more compartments are involved;
* Correction of varus or valgus.
* Willing to participate and return for follow-up study visits.

Exclusion Criteria:

* Vascular insufficiency
* Previous deep vein thrombosis and pulmonary embolism
* Previous osteotomy
* Previous patella fracture or surgery
* Previous healed tibia or femur fractures
* Previous joint replacement surgery

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mechanical Axis Alignment (Absolute Value Measured in Degrees) Using 3 Feet Long Leg Films | 3 Months Post-operative
  Femoral Valgus Angle, Tibial varus angle, Tibial slope, Femoral Flexsion/Extension angle, Implant Rotation

SECONDARY OUTCOMES:
Intraoperative Bleeding | Intra-operative
Operative time | During the procedure
Blood volume in suction drain | Post-operative Day 2
Hemoglobin level | Post-operative day1, 2, 3
WOMAC score | 6 weeks
WOMAC score | 3 Months
WOMAC score | 6 Months
WOMAC score | 1 year

OTHER OUTCOMES:
WOMAC Score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Phonthakorn Panichkul, MD, Principal Investigator — Thammasat University
Locations (1):
- Thammasat University Hospital., Pathum Thani, Changwat Pathum Thani, Thailand